CLINICAL TRIAL: NCT02027246
Title: Autologous Bone Marrow Mononuclear Cell Therapy for Spinal Cord Injury
Brief Title: Safety and Efficacy of Stem Cell Therapy in Spinal Cord Injury
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: Neurogen Brain and Spine Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NGBSI-05
Record Dates: First submitted 2013-12-18; First posted 2014-01-06 (Estimated); Last update posted 2018-10-25 (Actual); Status verified 2018-10

CONDITIONS: Spinal Cord Injury
Keywords: spinal cord injury; autologous bone marrow mononuclear cells; stem cell therapy
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Stem cell (Experimental): Autologous bone marrow mononuclear cell transplantation
  Interventions: Biological: Autologous bone marrow mononuclear cell transplantation

INTERVENTIONS:
Biological: Autologous bone marrow mononuclear cell transplantation — Bone marrow is aspirated by a standard procedure. Mononuclear cells are separated by density gradient method and then injected intrathecally by a standard lumbar puncture procedure

SUMMARY:
The aim of this study was to study the effect of stem cell therapy on common symptoms of spinal cord injury patients.

DETAILED DESCRIPTION:
Autologous bone marrow mononuclear cells are administered intrathecally by a standard procedure followed by standard rehabilitation therapy.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed cases of any type of chronic Spinal cord injury
* Age above 6 months

Exclusion Criteria:

* presence of acute infections such as Human immunodeficiency virus/ Hepatitis B Virus/ Hepatitis C Virus
* malignancies
* bleeding tendencies
* pneumonia
* renal failure
* severe liver dysfunction
* severe anemia [Hemoglobin < 8]
* any bone marrow disorder
* other acute medical conditions such as respiratory infection
* pregnancy and lactation

Ages: 8 Months to 63 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2008-12; Primary Completion 2012-08 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Change in clinical symptoms | 6 months
  clinical symptoms were assessed based on the observation of the experts

SECONDARY OUTCOMES:
Functional Independence Measure (FIM) | 6 months
  Functional Independence Measure (FIM) is a standard scale performed before and 6 months after the intervention to measure the functional ability of the patients.

CONTACTS AND LOCATIONS:
Overall Officials: Alok K Sharma, M.S., M.Ch, Principal Investigator — Neurogen Brain and Spine Institute
Locations (1):
- Neurogen brain and spine institute, Mumbai, Maharashtra, India

REFERENCES:
- [Background] Kumar AA, Kumar SR, Narayanan R, Arul K, Baskaran M. Autologous bone marrow derived mononuclear cell therapy for spinal cord injury: A phase I/II clinical safety and primary efficacy data. Exp Clin Transplant. 2009 Dec;7(4):241-8. PMID 20353375
- [Background] Yoshihara T, Ohta M, Itokazu Y, Matsumoto N, Dezawa M, Suzuki Y, Taguchi A, Watanabe Y, Adachi Y, Ikehara S, Sugimoto H, Ide C. Neuroprotective effect of bone marrow-derived mononuclear cells promoting functional recovery from spinal cord injury. J Neurotrauma. 2007 Jun;24(6):1026-36. doi: 10.1089/neu.2007.132R. PMID 17600518
- [Background] Sharma A, Gokulchandran N, Chopra G, Kulkarni P, Lohia M, Badhe P, Jacob VC. Administration of autologous bone marrow-derived mononuclear cells in children with incurable neurological disorders and injury is safe and improves their quality of life. Cell Transplant. 2012;21 Suppl 1:S79-90. doi: 10.3727/096368912X633798. PMID 22507683